CLINICAL TRIAL: NCT02001935
Title: Association Between CytochromeP4501A2(CYP1A2) and CytochromeP4502E1(CYP2E1) Gene Polymorphisms and Metabolism of Theophylline in a Chinese Population
Brief Title: Association Between CytochromeP4501A2 and CytochromeP4502E1 Gene Polymorphisms and Metabolism of Theophylline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 81302846
Record Dates: First submitted 2013-11-12; First posted 2013-12-05 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; theophylline; CYP1A2; CYP2E1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- theophylline (Other)
  Interventions: Drug: theophylline

INTERVENTIONS:
Drug: theophylline — After oral theophylline 200mg per day for two weeks,bood sample will be collected for determining plasma concentrations of theophylline and it's metabolites and the genotypes of CYP1A2 and CYP2E1

SUMMARY:
The aim of this study is to determine whether common CYP1A2 and CYP2E1 gene polymorphisms effect metabolism of theophylline in chronic obstructive pulmonary disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years,COPD patients, male or female;
* regularly visiting our hospital;
* taking a sustained-release preparation of theophylline continuously for at least 2 weeks

Exclusion Criteria:

* patients with renal or hepatic dysfunction;
* patients with congestive heart failure;
* patients with hypothyroidism or hyperthyroidism;
* patients currently taking drugs likely to affect theophylline metabolism or who had taken such drugs in the preceding week;
* patients with extreme obesity
* patients with very severe Chronic Obstructive Pulmonary Disease(COPD)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Theophylline clearance | Blood samples will be taken after receiving oral thoephylline for 14 days
  Theophylline and it's metabolite(1,3-dimethyluric) blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Wang Liqing, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China